CLINICAL TRIAL: NCT03883308
Title: The Influence of Multi-domain Cognitive Training on Large-scale Structural and Functional Brain Networks in MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Hadi Hosseini, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 120954; 5K25AG050759 (NIH)
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Treatment group will receive 6 months of online, computerized, multi-domain cognitive training at home.
  Interventions: Behavioral: Multi-domain cognitive training
- Active Control (Active Comparator): The Active Control group will receive 6 months of online, computerized cross-word puzzles at home using the same platform as for the Treatment group.
  Interventions: Behavioral: Cross-word puzzle training

INTERVENTIONS:
Behavioral: Multi-domain cognitive training — The cognitive exercises are designed to train executive functions and memory.
  Arms: Treatment
Behavioral: Cross-word puzzle training — The active control group will be asked to complete a variety of crossword puzzles using the same curriculum assigned to the TG group.
  Arms: Active Control

SUMMARY:
The purpose of this study is to integrate advanced computational techniques and multimodal neuroimaging methods to examine the potential effects of long-term, multi-domain, online, computerized cognitive training on large-scale structural and functional brain networks in older adults with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
This multilevel study will be comprised of a placebo controlled randomized controlled trial to test the effect of long-term (6 months), multi-domain, computerized cognitive training on large-scale structural and functional brain networks in individuals with MCI (age >= 65 years). Neuroimaging and neuropsychological data before and after intervention will be evaluated within and between groups to elucidate the trajectory of neuronal network improvements associated with training compared to typical MCI development. We will compare the outcomes between participants with MCI who receive structured cognitive training (treatment group: TG) with those who receive nonspecific computerized training activities (active controls: AC). The duration of intervention is 6 months. The focus of the study will be on individuals with amnestic MCI (single- or multi- domain). The study includes 30 MCI subjects in a treatment group (TG) and 30 matched MCI subjects in active control (AC) group. TG and AC participants will be evaluated at two time points: 1) baseline and 2) 6-month (post-training).

ELIGIBILITY:
Inclusion criteria:

* Cognitive concern by subject, informant or physician
* Impairment in memory domain (delayed recall of one paragraph from Logical Memory II subscale from Wechsler memory Scale - Revised with cutoff scores of <=8, <=4 and <=2 for 16, 8-15 and 0-7 years of education)
* Essentially normal functional activities
* Mini-Mental State Examination (MMSE) scores >=24
* Stability of permitted medications (e.g. cholinesterase inhibitors, hypertension medication, etc.) for at least two months.

Exclusion criteria:

* Any significant neurological condition including probable dementia, Parkinson's disease, Huntington's disease, multiple sclerosis, and brain tumor, among others.
* Presence of Axis I disorder
* Current use of psychoactive medications except for the permitted medications.
* Claustrophobia
* MRI contraindication
* Any significant systemic or unstable medical condition which could lead to difficulty complying with the protocol.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Executive function composite score | 6 months
  The primary behavioral outcome is executive function composite score that combines measures of working memory, inhibition, set-shifting, and fluency
Executive function network connectivity | 6 months
  The primary neuroimaging outcome is the interconnectivity of the frontal-striatal-parietal network.

SECONDARY OUTCOMES:
Memory function composite score | 6 months
  Memory function composite score that combines measures of auditory verbal learning and episodic memory
Medial temporal network connectivity | 6 months
  Regional interconnectivity and centrality in medial temporal network
White matter integrity in memory circuit | 6 months
  White matter integrity in posterior cingulate-medial temporal-frontal pathways

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Gozdas E, Avelar-Pereira B, Fingerhut H, Dacorro L, Jo B, Williams L, O'Hara R, Hosseini SMH. Long-term cognitive training enhances fluid cognition and brain connectivity in individuals with MCI. Transl Psychiatry. 2024 Oct 23;14(1):447. doi: 10.1038/s41398-024-03153-x. PMID 39443463